CLINICAL TRIAL: NCT05758844
Title: The Safe-line Technique as Additional Attempt to Mitigate Spinal Cord Ischemia After Endovascular Thoraco-abdominal Aneurysm Repair
Brief Title: The Safe-line Technique as Additional Attempt to Mitigate Spinal Cord Ischemia After Endovascular Exclusion of TAAA
Acronym: Safe-line-tech
Status: Recruiting | Type: Observational
Sponsor: University Hospital Padova (Other)
Responsible Party: Principal Investigator, Michele Piazza, Associate Professor, University Hospital Padova
Other Study IDs: Safe-line.1
Record Dates: First submitted 2023-01-30; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Thoracoabdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: safe-line technique — Safe-line approach

SUMMARY:
To assess safety and feasebility of the "safe-line" technique in a multicenter international collaboration.

DETAILED DESCRIPTION:
To assess safety and efficacy of a technique for temporary aneurysm sac re-perfusion (TASreP) after total endovascular exclusion of TAAA, using a guide-wire left into the aneurysm sac. The technique can be applied both in elective that urgent cases.

The guide-wire aim to be a "safe-line" for fast temporary trans-sealing aneurysm sac re-perfusion in case of SCI occurring in the early post-operative period (48-to 72h).

Before completing exclusion, from the percutaneous femoral access, a second buddy-wire (V-18 guidewire; Boston Scientific) is advanced and left posterior to the endograft into the aneurysmal sac; through the main guide-wire, the final aneurysm exclusion is completed with distal stent-graft deployment and the femoral access sealed with Proglide leaving in place the sole V.018 draped in a sterile fashion. In the case of SCI occurrence in the post-operative period up to 48-72 hrs, the trans-sealing V.18 "safe-line" can be rapidly exchanged with a 6F/65 cm long Destination cm guiding sheath (Terumo) and positioned into the aneurysmal sac; this can be connected to a 6F introducer from the contralateral femoral artery and the sac perfused in a retrograde fashion.

ELIGIBILITY:
Inclusion Criteria:

* Thoraco-abdominal aortic aneurysm including type I,II,III,IV and V.
* Pararenale aneurysm
* Thoracoabdominal aortic aneurysm Elective and Urgent, endovascular repair;
* Endovascular repair of any thoracoabdominal aortic condition

Exclusion Criteria:

-thoraco-abdominal aortic aneurysm open repair

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion of all patients treated for thoraco abdominal aortic aneurysm with endovascular repair and use of safe line technique
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-30 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | 7 days
  collect eventual complications (incidence of: 1- axis thrombosis; 2- microembolization; 3-hematoma)
Incidence of spinal cord ischemia improvement or resolution | 30 days
  collect all events that in case of post-operative (48-72hrs) spinal cord ischemia had symptoms mitigation (1-paraplegia improvement; 2 - paraplegia complete resolution)

CONTACTS AND LOCATIONS:
Locations (1):
- Vascular and Endovascular Clinic - Padova University, Padua, Italy

IPD SHARING:
Plan to Share IPD: Yes
With other partecipating centers